CLINICAL TRIAL: NCT06984991
Title: Factors Influencing Inadequacy in Rapid Onsite Evaluation of Ultrasound Guided Fine Needle Aspiration (FNA) Samples of Thyroid Nodules
Acronym: FNA inadequacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ramy Mohammed Ahmed, lecturer and consultant of radiology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: thyroid FNA
Record Dates: First submitted 2025-05-03; First posted 2025-05-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
Keywords: thyroid FNA
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thyroid FNA (Experimental): All FNAs will be performed by experienced radiologists (of 5-year experience in thyroid FNA procedures). Patients will be positioned comfortably, typically in a supine position with neck extension after putting a pillow under shoulders to fully expose the patient's neck to allow optimal access to the nodule. Ultrasound guidance using Logic E9 machine (GE Healthcare, Chicago, IL, USA) or Sonoscape X5 Portable Ultrasound machine with high-frequency linear array probes (3-12 MHz) will be used to visualize the nodule accurately and guide needle placement. 5ml syringe with 21G needle, 3ml syringe with 23G needle or 22G Quincke tip spinal needle will be used for FNA. Needle insertion will be directed either trans-isthmic or lateral cervical approach. Aspirations will be conducted at different angles and within different nodule regions using a to-and-fro motion till getting blood stain in the needle hub to obtain representative samples. Maximum number of four passes will be performed .
  Interventions: Diagnostic Test: fine needle aspiration

INTERVENTIONS:
Diagnostic Test: fine needle aspiration — Different needle sizes will be used in FNA sampling ; 5ml syringe with 21G needle, 3ml syringe with 23G needle or 22G Quincke tip spinal needle will be used for FNA. Needle insertion will be directed either trans-isthmic or lateral cervical approach. Aspirations will be conducted at different angles and within different nodule regions using a to-and-fro motion till getting blood stain in the needle hub to obtain representative samples. Maximum number of four passes will be performed within the nodule in a single session. Samples will be primarily obtained without suction via the capillary method. However, aspiration with suction will be applied if no aspirates could be obtained in the needle hub after routine capillary method. For mixed cystic solid lesions; FNA will be done from the solid component after aspiration of the cystic component

SUMMARY:
Thyroid nodules are a common clinical finding with a prevalence of around 50-67% in the general population using ultrasound examinations. Of these, malignancies account for 5-15% including the treatable papillary and follicular thyroid carcinomas and the rarer but more aggressive medullary and undifferentiated thyroid cancers.

Fine Needle Aspiration (FNA) is a relatively simple, cost-effective recommended standard diagnostic procedure with high sensitivity and specificity for the preoperative evaluation of benign and malignant thyroid nodules.

Cytopathology reports of thyroid FNA are categorized using a universal grading system, which helps to standardize reporting of diagnostic thyroid cytology results. In the non-diagnostic/unsatisfactory category (Bethesda I), ranging from 1% to 20% of samples, pathologists are unable to make a clinical diagnosis based on these samples due to an inadequate number of cells or difficulty in identifying cells. The estimated risk of malignancy in this category is 1-4 %, which usually managed by repeating FNA with increase in patient discomfort, procedural complications and medical costs.

There are few other prospective studies investigated the effect of needle size, and sampling technique on sample adequacy.

DETAILED DESCRIPTION:
Thyroid nodules are a common clinical finding with a prevalence of around 50-67% in the general population using ultrasound examinations. Of these, malignancies account for 5-15% including the treatable papillary and follicular thyroid carcinomas and the rarer but more aggressive medullary and undifferentiated thyroid cancers.

The American Thyroid Association has devised an algorithm "Thyroid Imaging Reporting and Data System (TI-RADS) for evaluation and management of thyroid nodules based on US pattern and size to recommend fine needle aspiration (FNA) cytology to minimize unnecessary FNAs/thyroid surgeries for nodules that are most likely benign and to avoid over-treating micropapillary thyroid carcinoma which is indolent. Fine Needle Aspiration (FNA) is a relatively simple, cost-effective recommended standard diagnostic procedure with high sensitivity and specificity for the preoperative evaluation of benign and malignant thyroid nodules.

Cytopathology reports of thyroid FNA are categorized using a universal grading system called The Bethesda System for Reporting Thyroid Cytopathology, which helps to standardize reporting of diagnostic thyroid cytology results [3]. In the non-diagnostic/unsatisfactory category (Bethesda I), ranging from 1% to 20% of samples, pathologists are unable to make a clinical diagnosis based on these samples due to an inadequate number of cells or difficulty in identifying cells. The estimated risk of malignancy in this category is 1-4 %, which usually managed by repeating FNA with increase in patient discomfort, procedural complications and medical costs.

Several retrospective and prospective studies investigated the factors associated with non-diagnostic samples rates, most of which focused on ultrasound guidance, the rapid on-site cytological evaluation and cystic components of the nodule. However, there are few other prospective studies investigated the other nodule characteristics, needle size, and sampling technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for FNA of thyroid nodules (TIRAD-3, 4 and 5 nodules).

Exclusion Criteria:

* History of thyroid ablation before FNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
rate of sample adequacy | Day 1
  Aspirated material will be expelled onto glass slides, which will be immediately fixed and stained for cytological analysis. Rapid On-Site Evaluation (ROSE) will be utilized to assess the sample adequacy during the procedure using the diff-quik (air-dried) slides, allowing for additional passes if necessary. In this situation, ROSE is not used for bedside diagnosis.
  An experienced pathologist reported the ical diagnosis/reporfinal cytologt only once the entire case (i.e. all of the slides) are reviewed according to the Bethesda criteria.:
  (I) nondiagnostic (ND) (fewer than six groups of well-visualized follicular cells, each group containing less than 10 well-preserved epithelial cells); (II) benign lesion; (III) atypia of undetermined significance/follicular lesion of undetermined significance (AUS/FLUS); (IV) follicular neoplasm/suspicious for follicular neoplasm (FN/SFN); (V) suspicious for malignancy; and (VI) malignancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sander CJ. Anaesthetic risk to tervuerens. Vet Rec. 1979 Nov 24;105(21):496. doi: 10.1136/vr.105.21.496. No abstract available. PMID 538881
- [Background] Cibas ES, Ali SZ. The Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2009 Nov;19(11):1159-65. doi: 10.1089/thy.2009.0274. PMID 19888858
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Moifo B, Moulion Tapouh JR, Dongmo Fomekong S, Djomou F, Manka'a Wankie E. Ultrasonographic prevalence and characteristics of non-palpable thyroid incidentalomas in a hospital-based population in a sub-Saharan country. BMC Med Imaging. 2017 Mar 4;17(1):21. doi: 10.1186/s12880-017-0194-8. PMID 28259145
- See also: Related Info — https://www.hopkinsmedicine.org/health/treatment-tests-and-therapies/thyroid-fine-needle-aspiration-biopsy